CLINICAL TRIAL: NCT02922712
Title: Evaluation of Clinical Efficacy and Safety of the Drug Nise (Nimesulide) in Complex Treatment of Patients With Osteoarthritis of the Knee and Hip Joints
Brief Title: Evaluation of the Efficacy and Safety of Nise 100 mg in the Management of Osteoarthrosis (Gonarthrosis)
Acronym: NISE-2013
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRL_RUS/MMD/2011/CT/NISE
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — nimesulide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NISE 100mg (Experimental): Nise 100mg given BD for 3 weeks
  Interventions: Drug: NISE

INTERVENTIONS:
Drug: NISE — Nise 200mg Max per day in 2 divided doses
  Other Names: Nimesulide

SUMMARY:
Study is conducted to evaluate safety and efficacy in patients with osteoarthritis

DETAILED DESCRIPTION:
Osteoarthritis is the most common disorders of the joints, which gives a page more than 10% of the world population aged over 45 years (Woolf A. D., Pfleger B., Bergman S., 2009). The main clinical manifestations of the disease are pain in the joints and a violation of their functions. Therefore, one of the first tasks in the therapeutic program, these patients will decrease and possible pain relief. Nesteroi dnye anti-inflammatory drugs (NSAIDs) are the main group of medicines drugs used in medical practice in lech th Research Institute of pain in patients with lesions of the musculoskeletal system. The basis of the therapeutic effect of the second of these drugs is the suppression of the activity of Fe p IU NTA cyclooxygenase (COX). Prichё m, the suppression of the activity of COX-2 isoenzyme involved in the synthesis of prostaglandins, induce the development of pain and PLAYBACK tion and provides anti-inflammatory effects of NSAIDs. B Blocking out of the enzyme COX-1, which controls the synthesis of prostaglandins, have cited a protective properties, leading to side effects of NSAIDs These so called nye formed the basis for the creation of new NSAIDs that can selectively inhibit COX-2 and m and mally affect COX. - 1.

Nimesulide is a selective inhibitor of cyclooxygenase -2 vnym with Sat and anced analgesic and anti-inflammatory effect, but also has antibradikinin, antihistamine and antioxidant activity of Stu(Nasonov EL, 1999, 2001).

ELIGIBILITY:
Inclusion Criteria:

* patients 40 years old and older with verified diagnosis of OA of the knee joints according to the criteria of American College of Rheumatology (АСR);
* radiologic abnormalities complying with I-III grades of Kellgren;
* pain syndrome not less than 40 points according to 100-point visual analogue scale (VAS).

Exclusion Criteria:

* A history of the patient within the last 5 years malignancy of any organ or system regardless of whether the treatment and is carried on this occasion elk.
* The presence of acute ulcer disease of the gastrointestinal tract that is, over several recent years.
* Any data on the bleeding from the upper gastrointestinal tract.
* Severe disease: uncontrolled hypertension, expression n naya cardiovascular failure, a pathology of the hematopoietic system, and mellitus type I, and others.
* The presence of other rheumatic diseases with the exception of teoartroza.
* Liver disease (cirrhosis, chronic hepatitis).
* Abnormal liver function (ALT, AST, bilirubin more than 1.5 times the upper limit of normal).
* Impaired renal function (blood creatinine more than 1.5 times higher than it's ver limit of normal).
* Anemia (g emoglobin more than 10 g / l less than the lower limit of normal).
* Treatment with corticosteroids (systemic reception), warfarin and other coumarin governmental produ d.
* Hypersensitivity to the analgesic and antipyretic Wed d stvam, NSAIDs, sulfonamides.
* Pregnancy and lactation.
* Alcohol and drug abuse history.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2011-03; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Mean Pain Intensity on VAS | From baseline to 3 week

CONTACTS AND LOCATIONS:
Overall Officials: Andrew E. Pihlak, MD, Principal Investigator — State Budgetary Institution of Higher Professional Education "A.I. Evdokimov Moscow State Medical Dental University" of the Ministry of Health of Russia

IPD SHARING:
Plan to Share IPD: Undecided